CLINICAL TRIAL: NCT00474448
Title: The Health-Related Quality of Life in Patients With Hereditary Multiple Exostoses
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: MHE Coalition (Unknown)
Responsible Party: Principal Investigator, Christine Alvarez, Principle Investigator, University of British Columbia
Other Study IDs: H07-00457
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2017-05

CONDITIONS: Exostoses, Multiple Hereditary
Keywords: Hereditary Multiple Exostoses; Survey; Quality of Life; Hereditary Multiple Exostoses,; also known as Multiple Hereditary Exostoses,; also known as Hereditary Multiple Osteochondromas
MeSH Terms: conditions — Exostoses, Multiple Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the health-related quality of life of subjects who have Hereditary Multiple Exostoses and to develop a disease specific quality of life survey. The investigators hypothesize that there are a wide range of quality of life experiences for patients with this syndrome.

DETAILED DESCRIPTION:
At the time of recruitment, subjects will be asked to indicate whether they would like to participate in a one-time survey, or are willing to participate in the initial survey plus two additional questionnaire administrations, thereafter, which will be used to develop the disease-specific quality of life (QOL) score. All participants will complete either the SF-36 survey (for adult HME subjects) or the CHQ PF (for parents of children with HME), as applicable, in addition to a blank form with categorical subheadings (such as recreation, social function, etc.), which they will use to address any issues not covered in the standardized questionnaire. Standardized questionnaires will be scored and analyzed. The items listed on the second form will be compiled and reapplied to subjects that indicated interest in extended participation in survey completion. Subjects will be asked to determine which items apply to them and to rank these applicable items in order of importance. The results from this will be used to develop a 30 question, disease-specific questionnaire. The final step will be to readminister this survey, in conjunction with the SF-36 or CHQ PF, and follow up, in two weeks, with a second administration of the aforementioned surveys, in order to test the variability and validity of the disease-specific, health-related, quality of life score.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with Hereditary Multiple Exostoses
* Adult patients or parents of child patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients or parents of child patients in British Columbia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
SF-36 score for adults and CHQ PF-50 for children | No time frame

CONTACTS AND LOCATIONS:
Overall Officials: Christine Alvarez, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada